CLINICAL TRIAL: NCT04911309
Title: Functional Exercise Intervention With Adolescents With Cerebral Palsy
Brief Title: Functional Exercise Training With Adolescents With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital Basel (Other)
Collaborators: Béatrice Ederer-Weber Stiftung (Unknown); Schweizerische Stiftung für das cerebral gelähmte Kind (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2020-02827; ks20Klaeusler
Record Dates: First submitted 2021-05-26; First posted 2021-06-03 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Palsy
Keywords: adolescents with cerebral palsy; functional exercise intervention; motor capability; motor capacity; gross motor function measure (GMFM-66)
MeSH Terms: conditions — Cerebral Palsy | interventions — Standard of Care; Therapeutics

STUDY DESIGN:
Intervention Model Description: This study is designed as a two-armed crossover intervention study with two intervention phases lasting 12 weeks each and three measurement points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: 12 weeks functional exercise training followed by standard therapy (Active Comparator): 12 weeks functional exercise training twice per week, each session lasting 60 min, additionally to standard therapy. Training sessions will be performed in a group-setting consisting of minimum 4 and maximum 8 participants and coached by experienced sport scientists with the supervision of a medical doctor. The exercises will be individually pants and constantly recorded in order to allow a progression over the course of the 12 week-period. The motor tasks and exercises will be tailored to individual capacity by experienced and trained sport scientists and coaches, therefore insuring the participants' safety and a continuous and progressive monitoring of training load.
  After 12 weeks the groups will switch the intervention method. Group 1 will therefore reassume their standard therapy for 12 weeks.
  Interventions: Other: functional exercise training; Other: standard therapy / treatment
- Group 2: 12 weeks standard therapy / treatment followed by 12 weeks functional exercise training (Active Comparator): 12 weeks standard therapy / treatment; the standard therapy group receives no additional exercise sessions. After 12 weeks the groups will switch the intervention method. Group 1 will therefore reassume their standard therapy for 12 weeks.
  After 12 weeks the groups will switch the intervention method. Group 2 will perform the same intervention which Group 1 received over the first course of 12 weeks.
  Interventions: Other: functional exercise training; Other: standard therapy / treatment

INTERVENTIONS:
Other: functional exercise training — 12 weeks functional exercise training twice per week, each session lasting 60 min
Other: standard therapy / treatment — 12 weeks standard therapy / treatment

SUMMARY:
This cross-over study analyzes a novel and inclusive approach in how therapy for adolescents with CP is administered, with the main goal of examining the effects of a functional exercise intervention on motor capability and motor capacity.

It is to investigate the effects of a functional movement-based exercise intervention in a group setting on motor capacity, motor capability and quality of life in adolescents with CP compared to standard therapy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a permanent disorder which affects the development of movement and posture. It causes activity limitation and is oftentimes accompanied by secondary musculoskeletal problems, disturbances of sensation, perception, cognition, communication and behavior.

In regard of the complex interplay between physical restrictions, motor disabilities, sedentary lifestyles and low participation in physical activity, an innovative exercise intervention study for adolescents with CP is intended in order to break the stated vicious cycle. This study aims at providing a novel and inclusive approach in how therapy for adolescents with CP is administered, with the main goal of examining the effects of a functional exercise intervention on motor capability and motor capacity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CP.
* Adolescents between 12 and 18 years of age.
* Gross Motor Functional Classification System (GMFCS): I-III.
* Cognitive abilities must include: Ability to actively engage in a training session of 60 min. duration; Ability to verbally or non-verbally communicate pain or discomfort; Ability to attend training, testing and follow-up sessions. All included participants are capable of making decisions on their own and no not show any signs of mental or cognitive limitations.

Exclusion Criteria:

* Any surgery or botulinum toxin treatment within 6 months prior to the start of the study or surgery/serial casting / botulinum toxin injection scheduled during the study period. Other medications can be continued as prescribed by the participants' physician.
* Known cardiovascular or pulmonary diseases that have not received medical clearance to participate in the physical exercise intervention.
* Uncontrolled seizures or epilepsy

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Function Measure-66 (GMFM-66) | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  assessment tool designed to measure changes in gross motor function over time in children and adolescents with CP. The test consist of the following five dimensions which span the spectrum of gross motor activities: a) lying and rolling; b) sitting; c) crawling and kneeling; d) standing; e) walking, running and jumping. Scores range from 0-3, higher scores denote better performance

SECONDARY OUTCOMES:
Change in height of participants | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  Change in height of participants will be measured in an upright standing position without shoes using a wall-mounted stadiometer
Change in body composition | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  Change in body composition will be measured by bioelectrical impedance analysis (BIA) using the InBody 270 (InBody Europe B.V., Eschorn, Germany) device
Change in clinical assessment | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  Clinical assessment will be performed for active ankle dorsiflexion, passive range of motion (RoM), spasticity according to the modified Ashworth/Bohannon scale (scale: 0-4). Tests resistance to passive movement about a joint with varying degrees of velocity. Scores range from 0-4, with 5 choices. A score of 1 indicates no resistance, and 5 indicates rigidity.
Change in muscle strength test (scale: 0-5) | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  Change in muscle strength test (scale: 0-5) : 0/5 = No visible muscle contraction. 5/5: Full strength
Change in arterial stiffness | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  Measurement of arterial stiffness using the oscillometric method. The mean values of three valid measurements will be calculated
Change in Six-minute walking test | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  The six-minute walking test will be performed between 2 lines set 20m apart. Participants will be instructed to walk as far as possible in 6 minutes.Total distance covered in six minutes as well as heart rate will be recorded.
Change in Handgrip Strength | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  Handgrip strength will be assessed using the Leonardo Mechanography GF®. Participants will be asked to hold their writing hand in a 90-degree angle and to squeeze the sensor as hard as possible for a total of 5 s. Participants will perform two valid measurements with 1 min rest in between. Peak strength in N as well as rate of force development (RFD) will be extracted.
Change in Bear Hug Carry | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  The bear hug carry will be performed carrying a medicine ball over a 100m distance. Two lines will be marked 20m apart and participants will be asked to walk the distance 5 times as fast as they can while holding the weighted ball in front of their chest. Participants at pre-measurement will be asked to carry the lightest ball (4 lbs). The same weight will be used in M2 as well as in M3 and the duration to walk the distance (in seconds) will be recorded. An additional test at M2 und M3 will be proposed, in which participants may choose an-other weight if they believe to be able to increase the load and repeat the test. This allows the measurement of individual increase in activity capacity. Weight and time will be recorded.
Change in Laying on the ground and standing up (burpees) | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  Individuals are to fully lay on the floor (hands, chest and feet) and stand or jump back up (full extension in hips and knees). The total number of repetitions over 60 seconds will be recorded
Change in Repeated Chair Rising Test (Box Squats): | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  The repeated chair rising test will be performed on a force plate (Leonardo Mechanography GF®, Novotec Medical GmbH, Pforzheim, Germany) with a 46cm high locked bench. Starting from a seated position, arms crossed in front of the chest, participants will perform five complete sit-to-stand cycles as fast as possible. Total time of the five repetitions as well as relative power and mean velocity for a cycle will be analyzed
Change in Isometric Mid-thigh pull | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  Isometric Mid-thigh pull (IMTP) is a multi-joint test which measures isometric force and rate of force development (RFD) in the back as well as lower body muscles and is strongly correlated to dynamic performance. Participants will be instructed to pull as fast and as hard as possible for a duration of 5 seconds
Change in Push Ups | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  The push up measures upper body strength (m. triceps brachii, m. pectoralis) and reflects the participants' ability to press and control their own body weight. For a full repetition, participants must start with their arms extended, touch the ground with their chest, and press back into an extended position. To find their 6 Repetition maximum (RM), participants will position their hands on a box with their feet on the floor. As in the squat depth test, depth of the boxes increase in a 10 cm increment. The lower the boxes, the more body weight is transferred on the upper body and must be pressed. Three minutes rest will be granted between trials to ensure complete recovery. The lowest box (or floor) on which 6 full repetitions can be performed will be noted. Box height and increase of active ROM will be analyzed.
Change in Medicine Ball over Bar Lift | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  This test measures the ability to lift and heave an object over an obstacle and allows a high trans-fer into daily life (i.e. lifting groceries onto a table or counter). Participants will lift a medicine ball from the ground and drop it over a bar installed in a rack at chest height as many times as possi-ble over 60 seconds, whereby testing personnel will roll the ball back in front of participants feet after every repetition. Weight of MB will be determined individually at M1 and corresponds to a 6 RM (whereby the lightest weight is a 4 lbs ball and the heaviest a 30 lbs medicine ball). Number of repetitions in the given time will be recorded. At M2 and M3, test will be repeated with the same medicine ball. Additionally, a new 6 RM will be determined and in the case of an increase in weight the test will be repeated with the new weight. Weight and number of repetitions will be recorded and increase in work capacity will be calculated.
Change in Seated sled pull | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  To assess participants' strength capacity in pulling strength, seated sled pulls will be performed. From a seated position, participants will pull a weighted sled over 20m using their upper body. Participants must pull the entire rope length (20m) without interruption in order for it to be counted as valid. The resistance (weight on the sled) will be increased in every round until failure (cannot pull rope or pull is interrupted). Weight and time of every round will be recorded.
Change in Maximum Power Output | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  Maximum power output and anaerobic capacity will be measured on an Assault Bike (Assault AirBike Classic ®, Ostfildern, Germany). Participants will perform a 1-minute all-out test. The resistance increases in line with rotations per minute (RPM). Participants will be instructed to go as hard as they can for the entire minute. Maximum heartrate and mean watt will be recorded and relative watt calculated to measure maximum power output.
Change in Accelerometry | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  In order to examine whether the intervention increases activity in daily life, patients will be asked to wear an Actigraph wGT3X-BT around their non-dominant wrist for 7 consecutive days and nights during each measuring phase. This triaxial accelerometer records intensity and duration of acceleration and converts the signals to "activity counts", allowing an analysis of duration and intensity of movement patterns during everyday life.
Change in instrumented gait analysis: temporospatial parameters | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  Change in instrumented gait analysis using a motion capture system. Participants will be asked to walk a distance of about 8 m at their self-selected speed. From the 3D gait data, the temporospatial parameters (cadence, stride length, and walking speed) can be calculated.
Change in instrumented gait analysis: Movement Analysis Profile (MAP) | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  Change in instrumented gait analysis using a motion capture system. Participants will be asked to walk a distance of about 8 m at their self-selected speed. From the 3D gait data, the Movement Analysis Profile (MAP) can be calculated.
Change in instrumented gait analysis: Profile Score (GPS) | at baseline (M1), at week 12 (M2: after intervention phase 1) and at week 24 (M3: after intervention phase 2)
  Change in instrumented gait analysis using a motion capture system. Participants will be asked to walk a distance of about 8 m at their self-selected speed. From the 3D gait data, the Gait Profile Score (GPS) can be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Elke Viehweger, Prof. Dr. med., Principal Investigator — Childrens University Hospital Basel (UKBB)
Locations (1):
- University Children's Hospital Basel, Basel, Switzerland